CLINICAL TRIAL: NCT06248931
Title: Valproate Versus Topiramate in Migraine, a Randomized Controlled Trial
Brief Title: Valproate Versus Topiramate in Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohamed G. zeinhom, MD, Dr., Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00000023988
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Migraine Disorders
Keywords: topiramate; valproate; migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Valproic Acid; Topiramate

STUDY DESIGN:
Intervention Model Description: We will assess The number of migraine days after three months of treatment, and the percentage of patients who achieved ≥ 50% reduction in the monthly headache days frequency compared to the baseline frequency (14). HIT-6 score reduction in each group after three months of treatment. The safety of treatment was evaluated by monitoring and documenting treatment-emergent adverse events (TEAE) in patients through regular follow-up procedures for three months.
Who Masked: Investigator, Outcomes Assessor
Masking Description: An independent statistician generated a blocked randomization sequence using computer-generated random numbers; participants received either valproate or topiramate from a specially trained and qualified nurse. We prepared Sequentially numbered opaque sealed envelopes and 600 labels for each drug labeled Drug A or B. According to the randomization chart, put them into envelopes numbered 1 to 600. Envelopes were attached to the patient's files. Patients were recruited sequentially and were given enrolment numbers starting from 1, which were mentioned on their files. Files with the same number as the patient enrolment number were opened and the patients were assigned to receive drugs A or B. Drug A included topiramate, and Drug B included valproate. The statistical analysis was performed by an independent statistician who did not know the treatment protocol of groups A or B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- valproate arm (Active Comparator): The arm will include 300 migraine patients diagnosed according to ICHD3-beta criteria. All patients will receive valproate 500-1000mg daily and Acetaminophen 500-1000 mg only in acute migraine attacks for 3 months. We will assess The change in migraine days per 28 days, the number of migraine days after three months of treatment, and the percentage of patients who achieved ≥ 50% reduction in the monthly headache days frequency compared to the baseline frequency (14). HIT-6 score reduction in each group after three months of treatment. The safety of valproate was evaluated by monitoring and documenting treatment-emergent adverse events (TEAE) in patients through regular follow-up procedures for three months.
  Interventions: Drug: Valproic acid
- topiramate arm (Active Comparator): The arm will include 300 migraine patients diagnosed according to ICHD3-beta criteria. All patients will receive topiramate 50-100mg daily and Acetaminophen 500-1000 mg only in acute migraine attacks for 3 months. We will assess The change in migraine days per 28 days, the number of migraine days after three months of treatment, and the percentage of patients who achieved ≥ 50% reduction in the monthly headache days frequency compared to the baseline frequency (14). HIT-6 score reduction in each group after three months of treatment. The safety of valproate was evaluated by monitoring and documenting treatment-emergent adverse events (TEAE) in patients through regular follow-up procedures for three months.
  Interventions: Drug: Topiramate 50 MG

INTERVENTIONS:
Drug: Valproic acid — The arm will include 300 migraine patients diagnosed according to ICHD3-beta criteria. All patients will receive valproate 500-1000 mg daily and Acetaminophen 500-1000 mg only in acute migraine attacks for 3 months. We will assess The change in migraine days per 28 days, the number of migraine days after three months of treatment, and the percentage of patients who achieved ≥ 50% reduction in the monthly headache days frequency compared to the baseline frequency (14). HIT-6 score reduction in each group after three months of treatment. The safety of valproate was evaluated by monitoring and documenting treatment-emergent adverse events (TEAE) in patients through regular follow-up procedures for three months.
  Other Names: group A
  Arms: valproate arm
Drug: Topiramate 50 MG — The arm will include 300 migraine patients diagnosed according to ICHD3-beta criteria. All patients will receive topiramate 50-100 mg daily and Acetaminophen 500-1000 mg only in acute migraine attacks for 3 months. We will assess The change in migraine days per 28 days, the number of migraine days after three months of treatment, and the percentage of patients who achieved ≥ 50% reduction in the monthly headache days frequency compared to the baseline frequency (14). HIT-6 score reduction in each group after three months of treatment. The safety of topiramate was evaluated by monitoring and documenting treatment-emergent adverse events (TEAE) in patients through regular follow-up procedures for three months.
  Other Names: group B
  Arms: topiramate arm

SUMMARY:
Investigators aim to compare the effect of valproate versus topiramate in migraine by assessing the reduction in MMD in each group, the percentage of patients who achieved ≥ 50% reduction in the monthly headache days frequency compared to the baseline frequency.

DETAILED DESCRIPTION:
Investigators will enroll 600 migraine patients who are diagnosed according to ICHD3-beta criteria in our study and will use a questionnaire to detect their demographic and clinical features (disease duration, attack frequency, and duration, pain intensity assessed by the visual analogic scale and we have two groups the first group will include 300 patients and will receive 500-1000mg valproate daily and Acetaminophen 500-1000 mg in acute attack, and the second group will receive topiramate100 mg per day and Acetaminophen 500-1000 mg in acute attack for at least three months. Investigators will assess The number of migraine days after three months of treatment and the percentage of patients who achieved ≥ 50% reduction in the monthly headache days frequency compared to the baseline frequency (14).. HIT-6 score reduction in each group after three months of treatment. The safety of treatment was evaluated by monitoring and documenting treatment-emergent adverse events (TEAE) in patients through regular follow-up procedures for three months.

ELIGIBILITY:
Inclusion Criteria:

Naive migraine patients, according to the International Classification of Headache Disorders 3rd edition, aged 18-75 years,

Exclusion Criteria

* Patients with major neurological disorders such as ( epilepsy, ischemic or hemorrhagic stroke, multiple sclerosis, mitochondrial diseases, brain tumors, and patients with essential tremors.
* Patients with major systemic diseases such as malignancy, collagen, liver, and renal diseases.
* Patients with cardiovascular diseases like hypertension (systolic blood pressure of more than 130 and/or diastolic blood pressure of more than 85 mm/Hg on at least three different occasions, diabetes (fasting plasma glucose level >126 mg/dl and/or a casual plasma glucose >200 mg/dl and/or HbA1C more than 6.5.
* Patients with valvular and ischemic heart diseases, bradycardia or heart blocks, congestive heart failure patients who received prophylactic treatment for migraine, patients with any contraindications to drugs used in the study Patients with topiramate or valproate contraindications.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
The percentage of patients who achieved ≥ 50% change in the monthly migraine days frequency compared to the baseline frequency. | 3 months
  We will assess The percentage of patients who achieved ≥ 50% change in the monthly headache days frequency compared to the baseline frequency in each group
The number of patients who discontinued treatment due to treatment-emergent adverse events. | 90 days
  The investigator will assess The number of patients who discontinued treatment due to treatment-emergent adverse events in each group after 3 months of treatment

SECONDARY OUTCOMES:
The severity of migraine attack on VAS score after three months of treatment | 3 months
  After three months of treatment, the investigators will assess the severity of migraine attacks on VAS scores.
  VAS is scale from one to ten where one is the least severe pain while ten is the severest pain
HIT-6 score change in each group after three months of treatment | 3 months
  The investigators assessed the absolute change in HIT6 score, the Headache Impact Test-6 (HIT-6) assessed the burden of headache in each group; the HIT-6 consists of six items: pain, social functioning, role functioning, vitality, cognitive functioning, and psychological distress, the patient answers each of the six related questions using one of the following five responses: "never", "rarely", "sometimes", "very often," or "always." These responses are summed to produce a total HIT-6 score that ranges from 36 to 78, where a higher score indicates a greater impact of headache on the daily life of the respondent. It has four impact grades: little-to-no impact (HIT-6 score: 36-49), moderate impact (HIT-6 score: 50-55), substantial impact (HIT-6 score: 56-59), and severe impact (HIT-6 score: 60-78)
Treatment safety was evaluated by monitoring treatment-emergent adverse events (TEAE) for three months. | 3 months
  The safety of treatment was evaluated by monitoring and documenting treatment-emergent adverse events (TEAE) in patients through regular follow-up procedures for three months.
The monthly migraine days per month | 30 days
  The investigators will assess the change in migraine days per month in each group.
The duration of migraine attack in hours after three months of treatment | 3 months
  After three months of treatment, the investigators will assess the duration of migraine attacks in hours in each group

CONTACTS AND LOCATIONS:
Overall Officials: mohamed G. Zeinhom, MD,PHD, Study Director — neurology department kafr el-sheikh university
Locations (1):
- Kafr Elsheikh University Hospital, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: No
All the data supporting this research's findings may be available from the principal investigator Mohamed G. Zeinhom upon reasonable request.

REFERENCES:
- [Result] Lipton RB, Scher AI, Kolodner K, Liberman J, Steiner TJ, Stewart WF. Migraine in the United States: epidemiology and patterns of health care use. Neurology. 2002 Mar 26;58(6):885-94. doi: 10.1212/wnl.58.6.885. PMID 11914403
- [Result] Lipton RB, Liberman JN, Kolodner KB, Bigal ME, Dowson A, Stewart WF. Migraine headache disability and health-related quality-of-life: a population-based case-control study from England. Cephalalgia. 2003 Jul;23(6):441-50. doi: 10.1046/j.1468-2982.2003.00546.x. PMID 12807523
- [Result] Mushet GR, Miller D, Clements B, Pait G, Gutterman DL. Impact of sumatriptan on workplace productivity, nonwork activities, and health-related quality of life among hospital employees with migraine. Headache. 1996 Mar;36(3):137-43. doi: 10.1046/j.1526-4610.1996.3603137.x. PMID 8984084
- [Derived] Zeinhom MG, Elsayed Khalil MF, Omar Youssif TY, Ali Daabis AM, Almoataz M, Refat HM, Mohamed Kamal Ebied AA, Atiaa Mohamed DM, Ismaiel M, Mohamed Kamel IF, Elballat AIE, Omar Akl AZ, Ahmed SR. Efficacy and tolerability of valproate versus topiramate in migraine prevention, a randomized controlled multi-center trial. J Clin Neurosci. 2025 May;135:111156. doi: 10.1016/j.jocn.2025.111156. Epub 2025 Feb 27. PMID 40020561